CLINICAL TRIAL: NCT05846555
Title: Comparison of Optic Nerve Sheath Diameter and Cerebral Regional Oxygen Saturation in Urological Surgery While Lithotomy Position
Brief Title: Optic Nerve Sheath Diameter in Urologic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Döndü Genc Moralar, Clinical Professor, Gaziosmanpasa Research and Education Hospital
Other Study IDs: 137/22
Record Dates: First submitted 2023-04-13; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Urological Manifestations; Anesthesia
Keywords: optic nerve sheath diameter; lithotomy position; near infrared spectrometer
MeSH Terms: conditions — Urological Manifestations | interventions — Urologic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- general anesthesia: patients observed under general anesthesia
  Interventions: Procedure: urologic surgery
- spinal anesthesia: patients observed under spinal anesthesia
  Interventions: Procedure: urologic surgery

INTERVENTIONS:
Procedure: urologic surgery — surgery

SUMMARY:
The investigators aimed to determine intracranial pressure changes during spinal and general anesthesia by using optic nerve sheath diameter and near infrared spectrometer in urologic surgery patients in lithotomy position. Also the investigators plan to evaluate to measure intrathoracic pressure effects to intracranial pressure.

DETAILED DESCRIPTION:
The patients will be divided into 2 groups as those who underwent general anesthesia and spinal anesthesia.Both groups at the specified times.

(The patient is supine for both groups before the start of the anesthesia procedure.) position T0, for group G, T1G 2 minutes after intubation, T1S 2 minutes after spinal anesthesia for group S, two T2, lithotomy 5 minutes after the lithotomy position for the group lithotomy to T3 30 minutes after the T4, T5 in PACU ) 60 minutes after optic nerve sheath diameter (OSC) values and lung assessment (LUS), cerebral cerebral palsy with Near-infrared spectroscopy (NIRS) oxygenation, mean arterial pressure, peripheral oxygen saturation, serum sodium, arterial carbon dioxide values and heart rate values will be recorded and significant statistical differences will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2-3, patients
* over 18 years of age who will undergo urological surgery

Exclusion Criteria:

* Existing disease that causes an increase in intracranial pressure
* Patients with optic nerve pathology,
* Ophthalmologic diseases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Urologic Surgery Patients
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-09-06 (Estimated); Study Completion 2023-12-05 (Estimated)

PRIMARY OUTCOMES:
intracranial pressure changes during Spinal and general anesthesia | position T0, for group G, T1G 2 minutes after intubation, T1S 2 minutes after spinal anesthesia for group S, two T2, lithotomy 5 minutes after the lithotomy position for the group lithotomy to T3 30 minutes after the T4, T5 in PACU ) 60 minutes after
  optic nerve sheat diameter as a predictor of intracranial pressure

CONTACTS AND LOCATIONS:
Overall Officials: zuhal çavuş, MD, Principal Investigator — gaziosmanpasa TREH
Locations (2):
- Turkey (Türkiye) (2):
  - Gaziosmanpaşa TREH, Istanbul, Gaziosmanpaşa
  - Gaziosmanpaşa TREH, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided